CLINICAL TRIAL: NCT03490643
Title: Temporomandibular Rahatsızlığın Postür ve Pedobarografik Ölçüm Sonuçları Ile İlişkisinin Araştırılması
Brief Title: An Investigation Of The Relationship Between Temporomandibular Disorder With Posture And Pedobarographic Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, PT. MSc. PhD (Candidate), Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 10840098-604.01.01-E.8466
Record Dates: First submitted 2018-03-25; First posted 2018-04-06 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-05

CONDITIONS: Temporomandibular Disorder
Keywords: Plantar Pressure Distribution; Posture; Posturescreen Mobile; RDC/TMD; TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMD Group (Other): people who has TMD
  Interventions: Other: Postural Analysis; Other: plantar pressure analysis
- Control Group (Other): individuals who dont have healthy temporomandibular joint
  Interventions: Other: Postural Analysis; Other: plantar pressure analysis

INTERVENTIONS:
Other: Postural Analysis — posture and plantar pressure analysis
Other: plantar pressure analysis — posture and plantar pressure analysis

SUMMARY:
The aim of the study is, to evaluate the whole body posture and plantar pressure distributions in individuals with Temporomandibular Disorder and also in people with healthy temporomandibular joints. A study group aged between 18-35 years, 30 patients, who were diagnosed with Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) who applied us with jaw pain and 30 healthy people at the same age range as a control group were included in the study. Both groups received global postural assessments by using PostureScreen Mobile® (PSM) program which is using four side photographs and the New York Posture Scale (NYPS). Static pedobarographic measurements were taken.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Temporomandibular Diseases
* clinical diagnosis of healthy temporomandibular joint

Exclusion Criteria:

* Trauma history
* Anatomic deformities and skeletal system fractures
* Orthopedic or rheumatic diseases diagnosed
* Pregnancy
* Having TMR treatment
* Being included in the physiotherapy program in the last 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
flexion and extension degree | 5 minutes
  degree
translation | 5 minutes
  cm

SECONDARY OUTCOMES:
plantar pressure distribution | 2 minutes
  kPa

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen, Principal Investigator — Medipol University; Zeliha Candan Algun, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)